CLINICAL TRIAL: NCT04137289
Title: A First-in-human Phase Ia/b, Open Label, Multicentre, Dose Escalation Study of BI 905711 in Patients With Advanced Gastrointestinal Cancers
Brief Title: A Study to Find a Safe and Effective Dose of BI 905711 in Patients With Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1412-0001; 2018-003268-29 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1a: Dose escalation (non randomised) Phase 1b: Dose expansion (randomised)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- BI 905711 0.02 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.02 milligram/kilogram (mg/kg) of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
  Interventions: Drug: BI 905711
- BI 905711 0.06 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.06 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
  Interventions: Drug: BI 905711
- BI 905711 0.2 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.2 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks.
  Interventions: Drug: BI 905711
- BI 905711 0.6 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.6 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
  Interventions: Drug: BI 905711
- BI 905711 0.6 mg/kg, QW (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.6 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every week for 3 weeks and then 1 week off (3 weeks on, 1 week off).
  Interventions: Drug: BI 905711
- BI 905711 1.2 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 1.2 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
  Interventions: Drug: BI 905711
- BI 905711 2.4 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 2.4 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
  Interventions: Drug: BI 905711
- BI 905711 3.6 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 3.6 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks.
  Interventions: Drug: BI 905711
- BI 905711 4.8 mg/kg, Q2W (Experimental): Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 4.8 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks.
  Interventions: Drug: BI 905711

INTERVENTIONS:
Drug: BI 905711 — BI 905711

SUMMARY:
Phase 1a - Explore safety and establish the maximum tolerated dose (MTD)/recommended dose levels for phase Ib expansion phase of BI 905711 based on the frequency of patients experiencing dose limiting toxicities (DLTs) during the MTD evaluation period. The MTD evaluation period is defined as the first two treatment cycles (from first dose administration until the day preceding the third dose administration or end of REP in case of discontinuation before start of Cycle 3).

Phase 1a - Explore pharmacokinetics/pharmacodynamics, and efficacy to guide the determination of a potentially effective dose range for phase Ib in the absence of MTD.

Phase 1b - Evaluate efficacy and safety of BI 905711 at a potentially effective dose range and determine the Recommended Phase 2 Dose (RP2D)

ELIGIBILITY:
Inclusion Criteria:

- a. Phase Ia (dose escalation only)

Histologically or cytologically confirmed, advanced unresectable or metastatic gastrointestinal cancers of following histologies:

* Colorectal adenocarcinoma
* Gastric adenocarcinoma
* Esophageal adenocarcinoma
* Pancreatic adenocarcinoma
* Cholangiocarcinoma and gallbladder carcinoma
* Small intestine adenocarcinoma b. Phase Ib (expansion phase)
* Histologically or cytologically confirmed, advanced unresectable or metastatic colorectal adenocarcinoma.

  * Patient who has failed all available conventional therapies known to confer clinical benefit for their disease based on local approved standards. For patients with colorectal cancer, prior treatment with regorafenib or TAS-102 is optional.
  * Phase Ia (dose escalation) only: Patient with either measurable or non-measurable/non-evaluable disease.
  * Phase Ia (expanded cohort) and Phase Ib (expansion phase) only: At least one target lesion that can be accurately measured per RECIST v.1.1
  * Availability and willingness to provide an archived tumor tissue specimen and undergo tumor biopsy before treatment. Pre-treatment fresh tumor biopsy collections for biomarker analyses are considered optional in phase Ia and mandatory in phase Ib. Only nonsignificant risk procedures per the investigator's judgment will be used to obtain any biopsies specified in this study. In case a fresh tumor biopsy cannot be obtained due to before mentioned reasons an archived tumor tissue specimen obtained within ≤6 months of screening must be submitted. In case the patient undergoes baseline tumor biopsy, an archived tumor tissue specimen must be submitted regardless of the date of collection.
  * Adequate hepatic, renal and bone marrow functions as defined by all of the below:
* Total bilirubin ≤ 1.5 x institutional Upper Level of Normal (ULN) (≤ 3 x institutional ULN for patient with Gilbert's syndrome)
* ALT and AST ≤2.5 x institutional ULN (≤5 x institutional ULN for patients with known liver metastases)
* Serum creatinine ≤1.5x institutional ULN. If creatinine is > 1.5 x ULN, patient is eligible if concurrent creatinine clearance ≥ 50 ml/min (>0.05 L/min) (measured or calculated by CKD-EPI formula or Japanese version of CKD-EPI formula for Japanese patients).
* ANC ≥ 1.0x 10^9/L (≥ 1.0 x 10^3/μL, ≥ 1,000/mm3)
* Platelets ≥ 100x10^9/ L (≥ 100 x 10^3/μL, ≥ 100 x 10^3/mm3)
* Hemoglobin (Hb) ≥8.5 g/dl, ≥ 85 g/L, or ≥ 5.3 mmol/L (without transfusion within previous week)
* Serum lipase ≤ 1.5 institutional ULN

  * Recovery from any adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 of previous anti-cancer therapies to baseline or CTCAE grade 1, except for alopecia CTCAE grade 2, sensory peripheral neuropathy CTCAE grade ≤ 2 or considered not clinically significant.
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
  * Life expectancy ≥ 3 months in the opinion of the investigator
  * Of legal adult age (according to local legislation) at screening
  * Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
  * Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

Exclusion Criteria:

* Previous systemic anti-cancer therapy within the specified timeframe from the last dose intake to the first dose of trial treatment as shown below:

  * Any non-investigational drug, including anti-angiogenic antibodies (bevacizumab or ramucirumab) and anti-EGFR antibodies (cetuximab or panitumumab), within 14 days.
  * Any investigational drug or other antibodies including immune checkpoint inhibitors, within 28 days.
* Radiation therapy within 4 weeks prior to start of treatment. However, palliative radiotherapy for symptomatic metastasis is allowed if completed within 2 weeks prior to start of treatment but must be discussed with the sponsor.
* Any serious concomitant disease or medical condition affecting compliance with Trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal (GI) tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator, would make the patient inappropriate for entry into the trial. Any history of stroke or myocardial infarction within 6 months prior to screening.
* Known pathological condition of GI tract, liver and pancreas, excluding the disease under study, that may interfere with assessment of drug safety or may increase the risk of toxicity:

  * inflammatory bowel disease
  * chronic pancreatitis
  * other serious GI pathological conditions by judgment of the investigator e.g. autoimmune disease with GI involvement, unexplained active diarrhea CTCAE grade ≥2 according to CTCAE v5.0.
* Known history of human immunodeficiency virus infection.
* Any of the following laboratory evidence of hepatitis virus infection. Test results obtained in routine diagnostics are acceptable if done within 14 days before the informed consent date:

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of HBc antibody together with HBV-DNA
  * Presence of hepatitis C RNA
* Active concomitant malignancies, other than the one treated in this trial.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes the patient an unreliable trial participant or unlikely to comply with the protocol requirements or not expected to complete the trial as scheduled.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial; female patients who do not agree to the interruption of breast feeding from the start of study treatment to within 30 days after the last study treatment.
* Presence of uncontrolled or symptomatic brain or subdural metastases. Inclusion of patients with brain metastases who have completed local therapy and are considered stable by the investigator, or with newly identified asymptomatic brain metastases at screening will be allowed. Use of corticosteroids is allowed if the dose was stable for at least 1 week before the baseline MRI.
* Patients who are under judicial protection and patients who are legally institutionalized
* Major surgery (major according to the investigator's assessment) performed within 3 weeks prior to treatment start or planned within 3 months after screening, e.g. hip replacement.
* Any of the following cardiac criteria:

  * Resting corrected QT interval (QTc) >470 msec
  * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block
  * Patients with an ejection fraction (EF) <50% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram, multi-gated acquisition scan). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
* Known hypersensitivity to the trial medication and/or its components i.e. polysorbate 20, sodium citrate, lysine hydrochloride, sucrose, citric acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Belgium (2):
  - Brussels - UNIV Saint-Luc, Brussels
  - UZ Leuven, Leuven
- China (2):
  - Beijing Cancer Hospital, Beijing
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
- France (4):
  - HOP Jean Minjoz, Besançon
  - CTR Leon Berard, Lyon
  - HOP la Milétrie, Poitiers
  - CTR Eugène Marquis, Rennes
- Universitätsklinikum Mannheim GmbH, Mannheim, Germany
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan
- Korea University Anam Hospital, Seoul, South Korea
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Garcia-Martinez JM, Wang S, Weishaeupl C, Wernitznig A, Chetta P, Pinto C, Ho J, Dutcher D, Gorman PN, Kroe-Barrett R, Rinnenthal J, Giragossian C, Impagnatiello MA, Tirapu I, Hilberg F, Kraut N, Pearson M, Kuenkele KP. Selective Tumor Cell Apoptosis and Tumor Regression in CDH17-Positive Colorectal Cancer Models using BI 905711, a Novel Liver-Sparing TRAILR2 Agonist. Mol Cancer Ther. 2021 Jan;20(1):96-108. doi: 10.1158/1535-7163.MCT-20-0253. Epub 2020 Oct 9. PMID 33037135
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objectives of this phase 1a/b, open-label, multicenter, dose escalation and dose expansion trial were to explore safety and establish maximum tolerated dose (MTD) of BI 905711 in patients with gastrointestinal cancers, as well as to explore pharmacokinetics, pharmacodynamics, and efficacy. Recruitment for the trial was discontinued during Phase 1b and no PDAC (pancreatic ductal adenocarcinoma) patients were enrolled as originally planned.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- BI 905711 0.02 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic gastrointestinal (GI) cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.02 milligram/kilogram (mg/kg) of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
- BI 905711 0.2 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.2 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
- BI 905711 0.6 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.6 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
- BI 905711 0.6 mg/kg, QW: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.6 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every week for 3 weeks and then 1 week off (3 weeks on, 1 week off).
- BI 905711 1.2 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 1.2 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
- BI 905711 2.4 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 2.4 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks. Participants in both the dose escalation and dose expansion phases at this dose were pooled together for baseline analysis.
- BI 905711 3.6 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 3.6 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
- BI 905711 4.8 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 4.8 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Period: Overall Study
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Started | 1 | 1 | 7 | 23 | 16 | 23 | 24 | 8 | 7
Treated in Phase 1a | 1 | 1 | 7 | 8 | 0 | 8 | 8 | 8 | 7
Treated in Phase 1b | 0 | 0 | 0 | 15 | 16 | 15 | 16 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 7 | 23 | 16 | 23 | 24 | 8 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Clinical disease progression | 0 | 0 | 0 | 4 | 4 | 2 | 5 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of clinical benefit | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Objective disease progression | 1 | 1 | 6 | 18 | 12 | 20 | 18 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. This TS was used for both safety and efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W | Total
Number analyzed (Participants) | 1 | 1 | 7 | 23 | 16 | 23 | 24 | 8 | 7 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 | 71.0 | 64.3 (6.7) | 56.0 (10.1) | 57.3 (10.5) | 57.7 (11.5) | 63.0 (10.9) | 64.9 (7.0) | 62.4 (6.8) | 59.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 9 | 7 | 16 | 10 | 2 | 2 | 47
  Male | 1 | 1 | 6 | 14 | 9 | 7 | 14 | 6 | 5 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0 | 8
  Not Hispanic or Latino | 1 | 1 | 7 | 19 | 14 | 18 | 19 | 8 | 7 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 0 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 2 | 1 | 2 | 4 | 2 | 2 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 4
  White | 0 | 0 | 5 | 17 | 13 | 18 | 18 | 5 | 4 | 80
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 0 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BI 905711 in Phase 1a
Description: Maximum tolerated dose (MTD) was defined as the highest dose with less than 25% risk of the true drug limiting dose (DLT) rate being equal to or above 33% during the MTD evaluation period. The MTD was to be considered reached if one of the following criteria was fulfilled: the posterior probability of the true DLT rate in the target interval (0.16, 0.33) of the MTD is above 0.5 or at least 15 patients have been treated in phase 1a, of which at least 6 were at the MTD.
Time Frame: From cycle 1 Day 1 until the second administration of study treatment (two 14-day treatment cycles).
Population: MTD evaluation set (MTDS): This included all patients in the treated set (TS) who were not replaced for the MTD determination. The MTDS was used for the primary analyses of drug limiting-toxicities (DLTs) and MTD determination. This analysis was carried out for participants in the Phase 1a part of trial.
Measure: Number; unit: milligram / kilogram (mg/kg)
Groups:
- BI 905711 0.02mg/kg - 4.8 mg/kg, Q2W: Comprises all dose cohorts during the dose escalation phase (phase 1a). Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration of 0.02mg/kg to 4.8 mg/kg of BI 905711 intravenously on Day 1 of each 14-day cycle.
Arm/Group | BI 905711 0.02mg/kg - 4.8 mg/kg, Q2W
Number analyzed (Participants) | 44
milligram / kilogram (mg/kg) | NA — The criteria for reaching the MTD were not fulfilled.

2. Primary Outcome: Number of Patients With Dose-limiting Toxicity (DLT) During the MTD Evaluation Period in Phase 1a
Description: Number of patients with dose-limiting toxicity (DLT) during the MTD evaluation period is reported.
Time Frame: From cycle 1 Day 1 until the day before cycle 3 Day 1 (two 14-day treatment cycles).
Population: MTD evaluation set (MTDS): This included all patients in the treated set (TS) who were not replaced for the MTD determination. The MTDS was used for the primary analyses of drug limiting-toxicities (DLTs) and MTD determination in Phase 1a.
Measure: Count of Participants; unit: Participants
Groups:
- BI 905711 0.2 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.2 milligram/kilogram (mg/kg) of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 6 | 8 | 7 | 8 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Confirmed Objective Response (OR) for Phase 1a and Phase 1b Combined
Description: Confirmed objective response (OR) as assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in patients with measurable disease is reported. This was defined as the best overall response of complete response (CR) or partial response (PR), where best overall response was the best response recorded from the start of the study treatment until the earliest of disease progression, death, or last evaluable tumor assessment and before start of subsequent anticancer therapy.
Time Frame: From the first administration of trial medication until the earliest of progressive disease (PD), death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, up to 48 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. The TS was used for both safety and efficacy analyses. While the protocol specified endpoints separately for Phase 1a/1b, final analysis of most endpoints (except pharmacokinetic and MTD endpoints) were based on the Treated set, with Phase 1a and 1b patients pooled, as seen here. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: Participants
Groups:
- BI 905711 0.02 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.02 milligram/ kilogram (mg/kg) of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 6 | 22 | 15 | 22 | 22 | 8 | 7
Participants | 0 [0 to 97.5] | 0 [0 to 97.5] | 0 [0 to 45.9] | 0 [0 to 15.4] | 0 [0 to 21.8] | 0 [0 to 15.4] | 0 [0 to 15.4] | 0 [0 to 36.9] | 0 [0 to 41.0]

4. Primary Outcome: Progression-free Survival (PFS)
Description: This was evaluated per RECIST 1.1 criteria for target lesions and assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. Overall response at each time point was evaluated by target lesion, non-target lesions and new lesions together, according to RECIST 1.1. Objective response (OR) was defined as best overall response of confirmed CR or confirmed PR according to RECIST 1.1.
Time Frame: From the first administration of trial medication until tumor progression or death, whichever occurred first, up to 48 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. This TS was used for both safety and efficacy analyses. Only participants with data were included in analysis and final analysis of PFS was based on the TS, with Phase 1a and Phase 1b patients pooled.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- BI 905711 1.2 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 1.2 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
- BI 905711 2.4 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 2.4 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 7 | 22 | 16 | 22 | 22 | 6 | 7
weeks | 6.29 [NA to NA] — Not calculable, as only one participant | 18.14 [NA to NA] — Not calculable, as only one participant | 5.71 [1.86 to 6.14] | 7.36 [5.29 to 12.00] | 7.43 [7.14 to 8.00] | 6.14 [4.57 to 8.00] | 7.14 [5.43 to 12.71] | 11.43 [4.86 to 20.14] | 7.43 [4.29 to 8.14]

5. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of BI 905711 During the First Cycle in Phase 1a
Description: Maximum measured plasma concentration (Cmax) of BI 905711 during the first cycle in phase 1a is reported.
Time Frame: Within 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after BI 905711 infusion in cycle 1.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Participants in the Phase 1a part were analyzed for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/ml)
Groups:
- BI 905711 0.6 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.6 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 4 | 8 | 5 | 8 | 8 | 7
nanograms/milliliter (ng/ml) | 306 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 492 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 2110 (16.1) | 6690 (18.4) | 11900 (29.5) | 26200 (24.3) | 40700 (22.5) | 61000 (26.9)

6. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of BI 905711 During the Third Cycle in Phase 1a
Description: Maximum measured plasma concentration (Cmax) of BI 905711 during the third cycle in phase 1a is reported.
Time Frame: Cycle 3: Within 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after BI 905711 infusion.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/ml)
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 4 | 6 | 8 | 6
nanograms/milliliter (ng/ml) | 336 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 497 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 2580 (17.5) | 7030 (20.9) | 10300 (44.8) | 31900 (26.4) | 47700 (23.9) | 50300 (32.1)

7. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-336) of BI 905711 During the First Cycle in Phase 1a
Description: Area under the concentration-time curve (AUC0-336) of BI 905711 during the first cycle in phase 1a is reported.
Time Frame: Within 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after BI 905711 infusion in cycle 1 .
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Due to premature discontinuation of the trial, no additional patients with pancreatic ductal adenocarcinoma were recruited. Only participants with available data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Groups:
- BI 905711 1.2 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 1.2 mg/kg of BI 905711 intravenously as a powder for solution for infusion, as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 0 | 1 | 4 | 7 | 5 | 8 | 8 | 7
hour*nanogram/milliliter (h*ng/mL) |  | 20000 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 97500 (39.5) | 391000 (50.1) | 872000 (39.8) | 1770000 (52.0) | 3330000 (22.3) | 4590000 (29.8)

8. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-336) of BI 905711 During the Third Cycle in Phase 1a
Description: Area under the concentration-time curve (AUC0-336) of BI 905711 during the third cycle in phase 1a is reported.
Time Frame: as for outcome 6
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Due to premature discontinuation of the trial, no additional patients with pancreatic ductal adenocarcinoma were recruited.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 0 | 1 | 3 | 6 | 4 | 4 | 7 | 5
hour*nanogram/milliliter (h*ng/mL) |  | 24500 (NA) — Geometric coefficient of variation could not be calculated for one subject. | 104000 (26.8) | 358000 (37.2) | 717000 (21.3) | 1990000 (76.3) | 3390000 (41.2) | 3990000 (63.3)

9. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of BI 905711 During the First Cycle in Phase 1b
Description: Maximum measured plasma concentration (Cmax) of BI 905711 during the first cycle in phase 1b is reported.
Time Frame: Within 5 minutes (min) before start of BI 905711 infusion and at 30 min, 7 hours (hrs), 24 hrs, 48 hrs, 168 hrs and 336 hrs after infusion in cycle 1. For 0.6 mg/kg QW only, there was no 336 hrs timepoint as the next drug was already given after 168 hrs.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This included all subjects in the treated set (TS) who provided at least one PK endpoint and were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/ml)
Arm/Group | BI 905711 0.6 mg/kg, QW | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W
Number analyzed (Participants) | 16 | 15 | 15 | 16
nanograms/milliliter (ng/ml) | 5740 (31.0) | 6150 (31.0) | 10700 (36.7) | 23100 (26.6)

10. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax) of BI 905711 During the Third Cycle in Phase 1b
Description: Maximum measured plasma concentration (Cmax) of BI 905711 during the third cycle in phase 1b is reported.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/ml)
Arm/Group | BI 905711 0.6 mg/kg, QW | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W
Number analyzed (Participants) | 12 | 10 | 11 | 12
nanograms/milliliter (ng/ml) | 5630 (28.0) | 6310 (47.8) | 13600 (39.5) | 23100 (20.9)

11. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-336) in Plasma of BI 905711 During the First Cycle in Phase 1b
Description: Area under the concentration-time curve (AUC0-336) in plasma of BI 905711 during the first cycle in phase 1b is reported. 11. The AUC calculation includes an extrapolation from 168 hrs to 336 hrs to account for the weekly dosing schedule.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | BI 905711 0.6 mg/kg, QW | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W
Number analyzed (Participants) | 14 | 15 | 15 | 16
hour*nanogram/milliliter (h*ng/mL) | 323000 (48.0) | 302000 (40.6) | 573000 (55.3) | 1460000 (50.0)

12. Secondary Outcome: Area Under the Concentration-time Curve (AUC0-336) in Plasma of BI 905711 During the Third Cycle in Phase 1b
Description: Area under the concentration-time curve (AUC0-336) in plasma of BI 905711 during the third cycle in phase 1b is reported. The AUC calculation includes an extrapolation from 168 hrs to 336 hrs to account for the weekly dosing schedule.
Time Frame: as for outcome 9
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | BI 905711 0.6 mg/kg, QW | BI 905711 0.6 mg/kg, Q2W | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W
Number analyzed (Participants) | 10 | 8 | 11 | 11
hour*nanogram/milliliter (h*ng/mL) | 354000 (42.9) | 339000 (48.1) | 571000 (78.9) | 1460000 (55.9)

13. Secondary Outcome: Number of Patients With Treatment-emergent Adverse Events (AEs)
Description: The number of patients with treatment-emergent adverse events (AEs) is reported, namely, all adverse events occurring between start of treatment and end of the residual effect period (REP). Adverse events that started before first drug intake and deteriorated under treatment were also considered as 'treatment-emergent'.
Time Frame: From start of treatment until the last dose of trial medication plus the residual effect period (REP), up to 358 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- BI 905711 4.8 mg/kg, Q2W: Comprises all dose cohorts during the dose escalation phase. Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration of 0.02mg/kg to 4.8 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 7 | 23 | 16 | 23 | 24 | 8 | 7
Participants | 1 | 1 | 5 | 22 | 16 | 23 | 20 | 8 | 7

14. Secondary Outcome: Maximum Percentage Change From Baseline in the Sum of Target Lesion Diameters
Description: Radiological (CT scan) tumor shrinkage, defined as the difference between the minimum post-baseline sum of longest diameters of target lesions and the baseline sum of the longest diameters of the same set of target lesions according to RECIST 1.1 is reported. Negative values indicate a reduction in the sum of target lesion diameters and positive values indicate an increase.
Time Frame: At baseline and every 8 weeks (± 7 days) until progression or start of further treatment for disease, up to 48 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. This TS was used for both safety and efficacy analyses. Only participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change in tumor diameter
Groups:
- BI 905711 4.8 mg/kg, Q2W: Comprises all dose cohorts during the dose escalation phase. Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration of 0.02mg/kg to 4.8 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 6 | 20 | 14 | 22 | 21 | 8 | 7
Percentage change in tumor diameter | 13.6 (NA) — Not calculable, as only 1 participant | -2.4 (NA) — Not calculable, as only 1 participant | 28.8 (13.85) | 20.8 (28.86) | 26.6 (26.43) | 34.3 (24.76) | 18.2 (25.90) | 19.3 (20.93) | 26.8 (23.02)

15. Secondary Outcome: Duration of Overall Response
Description: The duration of overall response was measured from the time measurement criteria were first met for complete response (CR) / partial response (PR) (whichever was first recorded) until the first date that recurrent or progression disease (PD) was objectively documented (taking as reference for PD the smallest measurements recorded in the study) according to RECIST 1.1.
Time Frame: From the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or PD is objectively documented, up to 48 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. This TS was used for both safety and efficacy analyses. Only participants with data were included in analysis and final analysis of overall response was based on the TS, with phase 1a and phase 1b patients pooled.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- BI 905711 4.8 mg/kg, Q2W: Comprises all dose cohorts during the dose escalation phase. Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration of 0.02mg/kg to 4.8 mg/kg of BI 905711 intravenously as a powder for solution for infusion, on Day 1 of each 14-day cycle.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 0 | 1 | 0 | 7 | 2 | 2 | 6 | 4 | 1
Days |  | 127.0 (NA) — Geometric coefficient of variation could not be calculated for one subject. |  | 170.3 (84.5) | 196.5 (119.5) | 87.0 (58.0) | 190.7 (78.7) | 90.5 (45.5) | 260.0 (NA) — Geometric coefficient of variation could not be calculated for one subject.

16. Secondary Outcome: Disease Control
Description: Disease control was defined as complete response (PR), partial response (PR), or stable disease according to RECIST 1.1 from the start of treatment until the earliest of progression disease (PD), death or last evaluable tumor assessment and before start of subsequent anti-cancer therapy. This endpoint analyzed the number of patients meeting this criterion.
Time Frame: From the start of treatment until the earliest of PD, death or last evaluable tumor assessment and before start of subsequent anti-cancer therapy, up to 48 weeks.
Population: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. This TS was used for both safety and efficacy analyses. Only participants with data were included in the analysis and final analysis of patients was based on the TS, with phase 1a and phase 1b patients pooled.
Measure: Count of Participants; unit: Participants
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
Number analyzed (Participants) | 1 | 1 | 6 | 22 | 15 | 22 | 22 | 8 | 7
Participants | 0 | 1 | 0 | 7 | 2 | 2 | 6 | 4 | 1

ADVERSE EVENTS:
Time Frame: Up to 358 days.
Description: Treated set (TS): This included all subjects who were dispensed study medication and were documented to have been treated with at least one dose of BI 905711. The TS was used for both safety and efficacy analyses.
Groups:
- BI 905711 0.02 mg/kg, Q2W: Patients with confirmed, advanced unresectable or metastatic GI cancers received a single administration (Cycle 1) and multiple administrations (Cycle 3) of 0.02 milligram/kilogram (mg/kg) of BI 905711 intravenously on Day 1 of each 14-day cycle treatment, once every two weeks.
Arm/Group | BI 905711 0.02 mg/kg, Q2W | BI 905711 0.06 mg/kg, Q2W | BI 905711 0.2 mg/kg, Q2W | BI 905711 0.6 mg/kg, Q2W | BI 905711 0.6 mg/kg, QW | BI 905711 1.2 mg/kg, Q2W | BI 905711 2.4 mg/kg, Q2W | BI 905711 3.6 mg/kg, Q2W | BI 905711 4.8 mg/kg, Q2W
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 5/7 | 15/23 | 6/16 | 15/23 | 11/24 | 7/8 | 4/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 2/7 | 14/23 | 4/16 | 7/23 | 10/24 | 2/8 | 1/7
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 5/7 | 22/23 | 16/16 | 23/23 | 19/24 | 7/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 905711 0.02 mg/kg, Q2W (N=1) | BI 905711 0.06 mg/kg, Q2W (N=1) | BI 905711 0.2 mg/kg, Q2W (N=7) | BI 905711 0.6 mg/kg, Q2W (N=23) | BI 905711 0.6 mg/kg, QW (N=16) | BI 905711 1.2 mg/kg, Q2W (N=23) | BI 905711 2.4 mg/kg, Q2W (N=24) | BI 905711 3.6 mg/kg, Q2W (N=8) | BI 905711 4.8 mg/kg, Q2W (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 905711 0.02 mg/kg, Q2W (N=1) | BI 905711 0.06 mg/kg, Q2W (N=1) | BI 905711 0.2 mg/kg, Q2W (N=7) | BI 905711 0.6 mg/kg, Q2W (N=23) | BI 905711 0.6 mg/kg, QW (N=16) | BI 905711 1.2 mg/kg, Q2W (N=23) | BI 905711 2.4 mg/kg, Q2W (N=24) | BI 905711 3.6 mg/kg, Q2W (N=8) | BI 905711 4.8 mg/kg, Q2W (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 6 | 3 | 3 | 5 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 6 | 2 | 6 | 5 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 3 | 4 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 4 | 4 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 5 | 11 | 4 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 4 | 6 | 5 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 5 | 1 | 5 | 3 | 1 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 3 | 2 | 5 | 3 | 2 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 3 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 4 | 0 | 5 | 3 | 0 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 0 | 1 | 4 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 4 | 0 | 4 | 4 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 5 | 0 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Carcinoembryonic antigen increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary occult blood positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 0 | 5 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 2 | 1 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 5 | 2 | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0 | 2 | 4 | 2 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Based on available preliminary data from Phase 1 clinical studies (1412-0001 and 1412-0003), the decision was made to terminate the BI 905711 (TRAILR2/CDH17) development program. This decision was not related to any safety concerns or unfavorable benefit/risk balance, but to the lack of predictive biomarkers and the limited efficacy, particularly in the context of the evolving treatment landscape for advanced colorectal cancer (CRC) and other gastrointestinal (GI) cancers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04137289/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04137289/SAP_001.pdf